CLINICAL TRIAL: NCT01285908
Title: Safety and Efficacy of Intravenous Norepinephrine for Orthostatic Hypotension
Brief Title: Intravenous Norepinephrine for Orthostatic Hypotension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110085; 11-N-0085
Record Dates: First submitted 2011-01-25; First posted 2011-01-28 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-09

CONDITIONS: Orthostatic Hypertension
Keywords: Baroreceptor; Norepinephrine; Orthostatic Hypotension; Sympathetic Nervous System; Blood Pressure
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baseline (No Intervention): Baseline values measured at various tilt angles, so that each participant may serve as their own control.
- Saline infusion (Placebo Comparator): Subjects received a saline IV infusion as a placebo, while measurements were taken at various tilt angles.
  Interventions: Drug: Intravenous Norepinephrine Infusion
- Norepinephrine Infusion (Active Comparator): Subjects were given an norepinephrine infusion at various tilt angles, while measurements were taken.
  Interventions: Drug: Intravenous Norepinephrine Infusion

INTERVENTIONS:
Drug: Intravenous Norepinephrine Infusion
  Arms: Norepinephrine Infusion; Saline infusion

SUMMARY:
Background:

- Orthostatic hypotension is a fall in blood pressure when standing up. Normally, a reflex action of the automatic nervous system makes blood vessels tighten when people stand up. The nervous system releases the chemical norepinephrine, which tightens blood vessels and keeps blood pressure in check. In orthostatic hypotension, the nervous system does not release enough norepinephrine when a person stands up, which can cause fainting or falling. Researchers are interested in determining whether norepinephrine given as a drug by vein can help maintain blood pressure during changes in body position.

Objectives:

- To determine whether intravenous norepinephrine can maintain blood pressure in people with orthostatic hypotension.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with orthostatic hypotension related to Parkinson's disease or pure autonomic failure.

Design:

* This study will require a 2-day inpatient admission to the NIH Clinical Center. The first day will involve laboratory evaluation and the second day will involve testing with norepinephrine. The second day requires an overnight stay.
* Participants will be screened with a medical history and physical examination, blood samples, and an electrocardiogram or echocardiogram.
* Participants who are on medications may be asked to taper or discontinue one or more medications for the purposes of this study. Participants may not take aspirin or any drugs that slow blood clotting for 7 days before study participation.
* Day 1: Participants will have a clear liquid breakfast, and will have a 1-hour baseline tilt table test to monitor blood flow, skin temperature, sweating, and blood pressure. Body temperature and breathing will also be monitored.
* Day 2: Participants will have a clear liquid breakfast, and will have a 2-hour tilt table test. Initial blood pressure readings will be taken, and an intravenous line will be placed. Participants will then receive norepinephrine or saline, followed by additional position changes of the tilt table to measure blood pressure differences before returning to the starting position. After about 10 minutes, the tilt table testing and infusion will be repeated with the other drug (saline or norepinephrine).
* Participants will be discharged 24 hours after the testing is complete.

DETAILED DESCRIPTION:
Objective:

Patients with chronic autonomic failure (CAF) often have disabling orthostatic hypotension (OH). In CAF, OH results from deficient baroreflex-mediated release of norepinephrine (NE) from sympathetic nerves. In patients with pure autonomic failure (PAF) or Parkinson disease (PD) with OH, cardiac and extra-cardiac noradrenergic denervation exacerbates effects of baroreflex failure. OH in CAF patients is often associated with supine hypertension, which can be severe. Drugs to treat OH worsen supine hypertension. Therefore, the combination of OH with supine hypertension poses a difficult therapeutic challenge. This protocol is a first step toward development of a prosthetic baroreceptor system to maintain blood pressure during orthostasis without worsening supine hypertension. In patients with PAF or PD+OH NE is infused i.v. at doses titrated individually to maintain blood pressure during head-up tilt at increasing angles from horizontal. Blood pressure is monitored continuously directly via an intra-arterial catheter. Because of the phenomenon of denervation supersensitivity, we anticipate that patients with OH associated with sympathetic noradrenergic denervation, as in PAF and PD, should be especially responsive to i.v. norepinephrine.

Study Population:

Patients with Parkinson disease and orthostatic hypotension or with pure autonomic failure.

Design:

This is a placebo controlled study that consists of two experimental days per participant. On a day before the day of norepinephrine (NE) infusion, the patient undergoes head-up tilting (typically at 15, 30, 45, and 60 degrees from horizontal) while blood pressure is monitored. Tilt angles are increased until the patient has orthostatic symptoms, systolic pressure decreases to less than 90 mm Hg, or systolic pressure decreases by more than 80 mm Hg. On the day of NE infusion patients, receive NE and placebo with the sequence of treatments randomized. If the patient has severe supine hypertension (more than 200 mm Hg systolic), then NE is infused beginning with the patient at whatever tilt angle is required for baseline pressure to be less than 200 mm Hg. NE is infused at doses titrated to keep directly recorded systolic blood pressure at or above the baseline value during exposure to higher tilt angles. When placebo is given, angles of tilt are increased until the patient has orthostatic symptoms, systolic pressure decreases to less than 90 mm Hg, or systolic pressure decreases by more than 80 mm Hg.

Outcome Measures:

The extent to which NE infusion can maintain blood pressure is tested by comparison of the fractional changes in systolic blood pressure at the same tilt angles during NE infusion vs. placebo infusion.

Primary:

1. Blood pressures (systolic, diastolic, mean)
2. Symptoms of orthostatic intolerance

Secondary:

1. Hemodynamics (e.g., total peripheral resistance)
2. Arterial plasma levels of norepinephrine and related neurochemicals

Comparison:

Patients undergo head-up tilt at the same angles to verify orthostatic hypotension if norepinephrine is not infused.

Participating Sites:

The study is done in the NIH Clinical Center in Bethesda, MD.

Contact Information:

The Principal Investigator is David S. Goldstein, MD PhD, Chief, Clinical Neurocardiology Section, CNP/DIR/NINDS/NIH, phone 301-496-2103, e-mail goldsteind@ninds.nih.gov. The contact for patient care coordination is Tereza Jenkins, phone 301-496-1115, e-mail jenkinst@ninds.nih.gov. The research contact (e.g., for database coordination) is Sandra Pechnik, phone 301-435-5166, e-mail pechniks@ninds.nih.gov.

ELIGIBILITY:
* INCLUSION CRITERIA:

A candidate subject is eligible for inclusion if he or she satisfies all of the following criteria:

Aged 18 years or over.

A confirmed diagnosis of neurogenic orthostatic hypotension related to Parkinson disease or pure autonomic failure.

Able to provide informed consent

EXCLUSION CRITERIA:

A candidate subject is ineligible for inclusion if he or she satisfies any of the following criteria:

Receiving medications expected to augment or attenuate blood pressure responses to i.v. norepinephrine (such as tricyclic antidepressants or alpha-adrenoceptor blockers).

Has heart block (unless a functioning cardiac pacemaker is in place or the patient is cleared by a cardiologist).

Raynaud's phenomenon or other findings in the medical history suggest a tendency to vasospasm.

History of myocardial infarction or current evidence of symptomatic congestive heart failure or symptomatic coronary ischemia.

Current evidence of ventricular arrhythmias or frequent premature ventricular contractions.

Renal failure.

History of mesenteric ischemia.

History of cerebrovascular ischemic disease, unless corrected (e.g., by stent).

Technical or medicinal limitations that obviate safe placement of arm intravenous and intra-arterial catheters for drug infusion and blood drawing. Examples of medicinal limitations are required daily aspirin ingestion and previously documented lidocaine allergy.

Pregnant or lactating or a female of child bearing potential who refuses to have a blood test for pregnancy. (Urine pregnancy tests can yield false-negative results, due to incorrect test preparation, urine that is too dilute, or interference by several medications. We have experience with the NIH Clinical Pathology Department not calling a urine test for pregnancy positive or negative because the urine was dilute. Serum pregnancy tests do not have these limitations.)

Unable to tolerate lying supine on a tilt table.

Closed angle glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Latour, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Polinsky RJ, Samaras GM, Kopin IJ. Sympathetic neural prosthesis for managing orthostatic hypotension. Lancet. 1983 Apr 23;1(8330):901-4. doi: 10.1016/s0140-6736(83)91329-6. PMID 6132222
- [Background] Oldenburg O, Mitchell A, Nurnberger J, Koeppen S, Erbel R, Philipp T, Kribben A. Ambulatory norepinephrine treatment of severe autonomic orthostatic hypotension. J Am Coll Cardiol. 2001 Jan;37(1):219-23. doi: 10.1016/s0735-1097(00)01062-7. PMID 11153742
- [Background] Goldstein DS, Horwitz D, Keiser HR, Polinsky RJ, Kopin IJ. Plasma l-[3H]norepinephrine, d-[14C]norepinephrine, and d,l-[3H]isoproterenol kinetics in essential hypertension. J Clin Invest. 1983 Nov;72(5):1748-58. doi: 10.1172/JCI111134. PMID 6630523
- [Background] Goldstein DS, Sewell L, Holmes C, Pechnik S, Diedrich A, Robertson D. Temporary elimination of orthostatic hypotension by norepinephrine infusion. Clin Auton Res. 2012 Dec;22(6):303-6. doi: 10.1007/s10286-012-0176-4. Epub 2012 Sep 16. PMID 22983778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through a NIH/NINDS screening protocol for Primary Chronic Autonomic Failure. Six subjects were enrolled during June 2011 to January 2012. Inclusion criteria required a confirmed diagnosis of neurogenic orthostatic hypotension related to Parkinson disease or pure autonomic failure.
Pre-assignment Details: Subjects underwent history and physical exam following consent. Subjects not meeting eligibility criteria were excluded prior to baseline testing. One subject was excluded prior to baseline testing due to recent stroke and one subject was terminated from the study during the testing phase due to examiner's inability to place an arterial line.
Groups:
- Baseline: Orthostatic hypotension was measured while lying flat (0 degrees) and at varying tilt angles (20, 40, and 60 degrees). Baseline measures included the following: blood pressure (systolic and diastolic), mean arterial pressure, heart rate, cardiac stroke volume, cardiac output, total peripheral resistance, plasma levels of norepinephrine and dihydroxyphenylglycol.
- Saline, Then Norepinephrine: Orthostatic hypotension was measured while lying flat (0 degrees) and at varying tilt angles (20, 40, and 60 degrees) under two separate conditions, i.e., first following IV administration of saline followed by IV administration of norepinephrine. Measures included the following: blood pressure (systolic and diastolic), mean arterial pressure, heart rate, cardiac stroke volume, cardiac output, total peripheral resistance, plasma levels of norepinephrine and dihydroxyphenylglycol.
- Norepinephrine, Then Saline: Orthostatic hypotension was measured while lying flat (0 degrees) and at varying tilt angles (20, 40, and 60 degrees) under two separate conditions, i.e., first following IV administration of norepinephrine followed by IV administration of saline. Measures included the following: blood pressure (systolic and diastolic), mean arterial pressure, heart rate, cardiac stroke volume, cardiac output, total peripheral resistance, plasma levels of norepinephrine and dihydroxyphenylglycol.
Period: Baseline Measurement
Arm/Group | Baseline | Saline, Then Norepinephrine | Norepinephrine, Then Saline
Started | 6 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — unable to insert catheter | 1 | 0 | 0
Not completed — History of stroke, exclusion criteria | 1 | 0 | 0
Not completed — unable to tolerate procedure | 1 | 0 | 0
Period: Treatment Crossover
Arm/Group | Baseline | Saline, Then Norepinephrine | Norepinephrine, Then Saline
Started | 0 | 2 (One subject in treatment crossover did not complete baseline testing as unable to complete tasks) | 2
Completed | 0 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are included for all subjects meeting eligibility criteria.
Groups:
- All Study Participants: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or Pure Autonomic Failure.
Arm/Group | All Study Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure (Systolic)
Description: The extent to which norepinephrine infusion maintains blood pressure, by comparison with the changes in systolic pressure at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: One subject was unable to tolerate tilting to 60 degrees following saline infusion and one subject was unable to tolerate tilting to 40 degrees following saline infusion; therefore the data for these subjects was not included in the saline condition.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with baseline measurements of systolic blood pressure taken at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of blood pressure taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of blood pressure taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
mm Hg
  Tilt Angle 0 | 156 (15) [141 to 171] | 158 (16) [142 to 174] | 179 (14) [165 to 193]
  Tilt Angle 20 | 148 (11) [137 to 159] | 149 (9) [140 to 158] | 173 (10) [163 to 183]
  Tilt Angle 40 | 131 (48) [83 to 179] | 128 (4) [124 to 132] | 167 (11) [156 to 178]
  Tilt Angle 60 | 112 (3) [109 to 115] | 120 (3) [117 to 123] | 175 (15) [160 to 190]

2. Primary Outcome: Blood Pressure (Diastolic)
Description: The extent to which norepinephrine infusion maintains blood pressure, by comparison with the changes in diastolic pressure at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure, with baseline measurements of diastolic blood pressure taken at varying tilt angles.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
mm Hg
  Tilt Angle 0 | 83 (7) [76 to 90] | 83 (2) [81 to 85] | 95 (6) [89 to 101]
  Tilt Angle 20 | 85 (6) [79 to 91] | 84 (3) [81 to 87] | 95 (4) [91 to 99]
  Tilt Angle 40 | 79 (4) [83 to 179] | 81 (4) [124 to 132] | 92 (5) [156 to 178]
  Tilt Angle 60 | 73 (3) [109 to 115] | 80 (4) [117 to 123] | 98 (7) [160 to 190]

3. Secondary Outcome: Heart Rate
Description: The extent to which norepinephrine infusion affects heart rate, by comparison of beat-to-beat heart rate at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with baseline measurements of heart rate taken at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of heart rate taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of heart rate taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
bpm
  Tilt Angle 0 | 62 (4) [58 to 66] | 55 (8) [47 to 63] | 58 (5) [53 to 63]
  Tilt Angle 20 | 57 (2) [55 to 59] | 56 (3) [53 to 59] | 60 (4) [56 to 64]
  Tilt Angle 40 | 55 (3) [52 to 58] | 58 (3) [55 to 61] | 59 (4) [55 to 63]
  Tilt Angle 60 | 65 (3) [62 to 68] | 63 (4) [59 to 67] | 63 (2) [61 to 65]

4. Secondary Outcome: Cardiac Stroke Volume
Description: The extent to which norepinephrine infusion affects cardiac stroke volume, by comparison of cardiac stroke volume at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure, with baseline measurements of cardiac stroke volume taken at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of cardiac stroke volume taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of cardiac stroke volume taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
mL
  Tilt Angle 0 | 76 (15) | 66 (20) | 83 (13)
  Tilt Angle 20 | 70 (15) | 62 (20) | 82 (13)
  Tilt Angle 40 | 62 (13) | 56 (18) | 76 (11)
  Tilt Angle 60 | 52 (5) | 50 (14) | 67 (12)

5. Primary Outcome: Blood Pressure (Mean)
Description: The extent to which norepinephrine infusion maintains average blood pressure, by comparison with the fractional changes in blood pressure at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure, with baseline measurements of average blood pressure taken at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of average blood pressure taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of average blood pressure taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
mm Hg
  Tilt Angle 0 | 107 (10) | 108 (7) | 123 (9)
  Tilt Angle 20 | 106 (8) | 106 (5) | 121 (6)
  Tilt Angle 40 | 96 (45) | 97 (4) | 116 (7)
  Tilt Angle 60 | 86 (3) | 93 (3) | 124 (9)

6. Secondary Outcome: Cardiac Output
Description: The extent to which norepinephrine infusion affects cardiac output, by comparison of cardiac output at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure, with baseline measurements of cardiac output taken at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of cardiac output taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of cardiac output taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
L/min
  Tilt Angle 0 | 4.6 (0.6) | 3.8 (1.6) | 4.9 (1.0)
  Tilt Angle 20 | 3.9 (0.7) | 3.5 (1.3) | 5.1 (1.0)
  Tilt Angle 40 | 3.4 (0.5) | 3.3 (1.2) | 4.6 (0.9)
  Tilt Angle 60 | 3.4 (0.4) | 3.2 (1.1) | 4.2 (0.8)

7. Secondary Outcome: Total Peripheral Resistance
Description: The extent to which norepinephrine infusion affected total peripheral resistance, by comparison of total peripheral resistance at varying tilt angles during baseline and saline infusion.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg/(min/L)
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure, with baseline measurements of total peripheral resistance taken at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of total peripheral resistance taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of total peripheral resistance taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
mmHg/(min/L)
  Tilt Angle 0 | 22.4 (1.6) [20.8 to 24.0] | 34 (16) [18 to 50] | 27 (6) [21 to 33]
  Tilt Angle 20 | 26.9 (3.1) [23.8 to 30] | 33 (14) [19 to 47] | 26 (7) [19 to 33]
  Tilt Angle 40 | 27.7 (3.5) [24.2 to 31.2] | 32 (13) [19 to 45] | 28 (7) [21 to 35]
  Tilt Angle 60 | 24.5 (2.8) [21.7 to 27.3] | 30 (9) [21 to 39] | 31 (6) [25 to 37]

8. Secondary Outcome: Arterial Plasma Levels of Norepinephrine
Description: Plasma levels of norepinephrine are obtained from blood samples via IV catheter.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with baseline measurements of plasma levels of norepinephrine at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of plasma levels of norepinephrine taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of plasma levels of norepinephrine taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
nmol/L
  Tilt Angle 0 | 0.78 (0.29) [.49 to 1.07] | 0.82 (0.33) [.49 to 1.15] | 0.73 (0.22) [.51 to .95]
  Tilt Angle 20 | 0.89 (0.34) [.55 to 1.23] | 0.65 (0.22) [.43 to 0.87] | 1.99 (0.67) [1.32 to 2.66]
  Tilt Angle 40 | 1.04 (0.4) [.64 to 1.44] | 0.97 (0.39) [.58 to 1.36] | 3.73 (0.94) [2.79 to 4.67]
  Tilt Angle 60 | 1.3 (0.48) [.82 to 1.78] | 2.32 (0.02) [2.3 to 2.34] | 7.83 (1.4) [6.43 to 9.23]

9. Secondary Outcome: Arterial Plasma Levels of Dihydroxyphenylglycol (DHPG)
Description: Plasma levels of dihydroxyphenylglycol are obtained from blood samples via IV catheter.
Time Frame: 2 experimental days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Baseline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure, with baseline measurements of plasma levels of dihydroxyphenylglycol at varying tilt angles.
- Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of plasma levels of dihydroxyphenylglycol taken at varying tilt angles following a saline infusion.
- Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements of plasma levels of dihydroxyphenylglycol taken at varying tilt angles following a norepinephrine infusion.
Arm/Group | Baseline | Saline | Norepinephrine
Number analyzed (Participants) | 3 | 2 | 4
nmol/L
  Tilt Angle 0 | 3.42 (0.26) | 4.01 (0.32) | 4.07 (0.40)
  Tilt Angle 20 | 3.44 (0.22) | 3.97 (0.28) | 4.05 (0.34)
  Tilt Angle 40 | 3.82 (0.46) | 4.18 (0.30) | 4.12 (0.45)
  Tilt Angle 60 | 4.39 (0.56) | 5.00 (0.33) | 4.47 (0.52)

ADVERSE EVENTS:
Groups:
- Baseline: The participants are patients with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with baseline measurements of BP at varying tilt angles.
- Saline, Then Norepinephrine: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements taken at varying tilt angles under two separate conditions, i.e., following IV administration of saline, followed by IV administration of norepinephrine.
- Norepinephrine, Then Saline: The participants are subjects with neurogenic orthostatic hypotension associated with Parkinson disease or pure autonomic failure with measurements taken at varying tilt angles under two separate conditions, i.e., following IV administration of norepinephrine, followed by IV administration of saline.
Arm/Group | Baseline | Saline, Then Norepinephrine | Norepinephrine, Then Saline
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 0/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (N=6) | Saline, Then Norepinephrine (N=2) | Norepinephrine, Then Saline (N=2)
Eccymoses (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Ecchymoses in the arms after failed attempts to place brachial and radial arterial catheters

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No